CLINICAL TRIAL: NCT03300947
Title: Psilocybin for Treatment of Obsessive Compulsive Disorder
Acronym: PSILOCD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Francisco A Moreno, Associate Vice President, Diversity and Inclusion; Professor, Psychiatry, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1707613822
Record Dates: First submitted 2017-09-14; First posted 2017-10-04 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Obsessive-compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psilocybin; Lorazepam

STUDY DESIGN:
Intervention Model Description: All participants will be randomly assigned to administration of low dose (100 µg/kg) psilocybin, High dose (300 µg/kg) psilocybin, or Lorazepam (1 mg). Eight different sessions divided in two phases will ensure all subjects are exposed to psilocybin at some point during the study in a blinded fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase One: Double blind (both participant AND researchers (In room Care Provider, Investigators, Blinded Outcomes Assessor) Phase Two: Single blind (Participant and Blinded Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High-dose Psilocybin (Experimental): Psilocybin 300 mcg/kg once per week, every week, for 8 weeks
  Interventions: Drug: Psilocybin 300 mcg/kg
- High- or Low-dose Psilocybin (Experimental): Psilocybin 100 mcg/kg or psilocybin 300 mcg/kg once per week, every week, for 8 weeks
  Interventions: Drug: Psilocybin 100 mcg/kg; Drug: Psilocybin 300 mcg/kg
- High-dose Psilocybin or Lorazepam (Placebo Comparator): Psilocybin 300 mcg/kg or Lorazepam 1 mg once per week, every week, for 8 weeks
  Interventions: Drug: Psilocybin 300 mcg/kg; Drug: Lorazepam 1 mg

INTERVENTIONS:
Drug: Psilocybin 100 mcg/kg — Psilocybin belongs to the class of hallucinogen or psychedelic drugs. It is one of the major psychoactive components in mushrooms of the Psilocybe genus ("magic mushrooms").
  Other Names: Psilocybine, "magic mushrooms"
  Arms: High- or Low-dose Psilocybin
Drug: Psilocybin 300 mcg/kg — Psilocybin belongs to the class of hallucinogen or psychedelic drugs. It is one of the major psychoactive components in mushrooms of the Psilocybe genus ("magic mushrooms").
  Other Names: Psilocybine, "magic mushrooms"
Drug: Lorazepam 1 mg — A medication used to treat anxiety belonging to a class of drugs known as benzodiazepines, which act on the central nervous system to produce a calming effect. This drug works by enhancing the effects of a certain natural chemical in the body (GABA).
  Other Names: Ativan, Intensol
  Arms: High-dose Psilocybin or Lorazepam

SUMMARY:
This study will evaluate whether psilocybin, a hallucinogenic drug, improves symptoms of obsessive compulsive disorder (OCD), whether it is safely tolerated as treatment of OCD, and will investigate the mechanisms by which it works.

DETAILED DESCRIPTION:
The study seeks to improve our ability to treat and improve the lives of people who have obsessive-compulsive disorder (OCD) by exploring the benefits of psilocybin, a mind-altering drug that changes activity in brain areas believed to be involved in OCD. Anecdotal reports and results from previous research support this idea. This two-phase study will enroll patients with symptomatic OCD who are not taking mind-altering medications or street drugs.

During Phase One, neither participants nor the investigators will know which drugs or doses are administered. This information will be available if it is medically necessary to reveal which drugs and doses were administered. Five subjects in each group will receive study drug a total of four times, separated by one week. During Phase Two, participants will not know which drugs or doses they receive, but the investigators will know. All participants will receive psilocybin at some point during study participation.

Participants will be randomly assigned to one of the following groups:

1. Low dose (100 µg/kg) psilocybin,
2. High dose (300 µg/kg) psilocybin, or
3. Lorazepam (1 mg), a calming medication. Lorazepam is used often for anxiety and will be used to mask which drug participants receive.

Participants will spend approximately 12 hours at the research site under observation during each visit, until they are free of the mind-altering effects of the drug and are determined by the psychiatrist to be safe to go home accompanied by a responsible adult. The effects of low versus high doses, and the additive effects of repeated doses will be analyzed and will be compared to the effects of lorazepam.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe OCD (DSM-5) after diagnostic interview using the Structured Clinical Interview for DSM-5 Research Version (SCID-R).
* Failed at least one adequate attempted routine care treatment.
* Considered safe for independent living

Exclusion Criteria:

* Concurrent psychosis, active substance use disorder, or a personal history of psychosis.
* Medical illness based on physical examination and routine blood testing that may complicate cardiovascular safety or drug metabolism or excretion, such as uncontrolled hypertension, severe cardiac disease, or kidney or liver failure.
* Unstable Chronic Obstructive Pulmonary Disease (COPD) or severe sleep apnea
* Psychiatric comorbidity that may represent an acute risk to their own or others' safety.
* Subjects may not be using antidepressant medication for OCD for at least two weeks before receiving study drug, and they cannot require any sedative, narcotic, or neuroleptic medications on a regular basis. Any of these medications they have taken should have been stopped long enough in the past to allow for their elimination and safe withdrawal prior to starting administration of the study drug. The specific time required will be dependent on the medication the patient was previously receiving.
* Women who are pregnant, breastfeeding, or unwilling/unable to practice medically acceptable birth control during the study.
* Allergy to lorazepam.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Treatment-phase effects on Obsessive-Compulsive symptom severity | weekly Y-BOCS rating prior to ingestion of study drug on Week 1 through 8, and week 9 (follow up week 1)
  Prospective Assessment of YBOCS (Yale-Brown Obsessive Compulsive Scale) score comparing each psilocybin dose and active placebo (Lorazepam).

SECONDARY OUTCOMES:
Acute Incidence of Treatment Emergent Adverse Events | At 0, and 24 hours after blinded medication ingestion
  Prospective active inquiry of adverse events with the SAFTEE-GI (Systematic Assessment For Treatment Emergent Events-General Inquiry) comparing each psilocybin dose and active placebo (Lorazepam)
Duration of Effects on Obsessive-Compulsive symptom severity | Follow-up assessments will be conducted weekly over the phone weekly (± 3 days) for one month after last dose, monthly (± 7 days) for three months beginning 28 days after last dose, and then once at 6 months after last dose (± 7 days).
  Prospective Naturalistic Assessment of YBOCS (Yale-Brown Obsessive Compulsive Scale) after repeated administration of study drug.
Long Term Incidence and Duration of Treatment Emergent Psychiatric Adverse Events | Follow-up assessments will be conducted weekly over the phone (± 3 days) for one month after last dose, monthly (± 7 days) for three months beginning 28 days after last dose, and then once at 6 months after last dose (± 7 days).
  Prospective Assessment with SCID-I (Structured Clinical Interview for DSM-5 Disorders) psychotic screening tool will assess for onset of psychopathology or hallucinogen induced disorders after repeated use.
Changes in the magnitude of Error Related Negativity (an electroencephalographic biomarker of OCD) assessed by Error-related negativity (voltage) and mid-frontal theta power (time-frequency approach) | Baseline, and 9-10 hours after ingestion of study dose 1, 4, and 8.
  Prospective Assessment of Error Related brain activity comparing each psilocybin dose and active placebo (Lorazepam).
Prospective Self-Assessment of Depression Symptoms | Baseline, 24 hours after each dose during 8 week active phase, and during the follow-up phase (weekly for one month after last dose, monthly for three months beginning 28 days after last dose, and then once at 6 months after last dose.
  Prospective Assessment of Quick Inventory of Depressive Symptomatology (QIDS) Score comparing each psilocybin dose and active placebo (Lorazepam).
Prospective Clinician-Rated Assessment of Depression Symptoms | Baseline, 4 weeks, 8 weeks, and during the follow-up phase (weekly for one month after last dose, monthly for three months beginning 28 days after last dose, and then once at 6 months after last dose
  Prospective Assessment of Montgomery-Asberg Depression Rating Scale (MADRS) Score comparing each psilocybin dose and active placebo (Lorazepam).
Changes in functional connectivity: 1) between the Caudate Nucleus (CN) and Orbital Frontal Cortex (OFC); 2) within the default mode network (DMN). | Imaging at baseline, and 9-10 hours post ingestion on weeks 1, 4, and 8. YBOCS at baseline and 8 hours after ingestion at weeks 1, 4, and 8.
  Prospective Assessment of Functional Connectivity in CN and OFC and in DMN comparing each psilocybin dose and active placebo (Lorazepam). Also examining whether magnitude of symptom reduction is related to changes in functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A. Moreno, MD, Principal Investigator — Professor of Psychiatry and Associate Vice President, Diversity and Inclusion
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moreno FA, Wiegand CB, Taitano EK, Delgado PL. Safety, tolerability, and efficacy of psilocybin in 9 patients with obsessive-compulsive disorder. J Clin Psychiatry. 2006 Nov;67(11):1735-40. doi: 10.4088/jcp.v67n1110. PMID 17196053
- See also: PubMed Abstract Link — https://www.ncbi.nlm.nih.gov/pubmed/?term=17196053